CLINICAL TRIAL: NCT05906004
Title: Post-Market Clinical Follow-up (PMCF) Study of the Pitch-Patch for the Augmentation or Reinforcement of the Rotator Cuff
Status: Not yet recruiting | Type: Observational
Sponsor: Xiros Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CRE 031
Record Dates: First submitted 2023-05-25; First posted 2023-06-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Rotator Cuff Tear; Rotator Cuff Tears; Rotator Cuff Tears of the Shoulder; Rotator Cuff Injuries
Keywords: Rotator Cuff Reinforcement; Rotator Cuff Repair; Pitch-Patch; Xiros; Rotator Cuff Augmentation
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pitch-Patch — Pitch-Patch device used for rotator cuff augmentation/ reinforcement.

SUMMARY:
This is a clinical investigation study. It will verify the long-term safety and performance of the Pitch-Patch when implanted to reinforce partially repairable rotator cuff tears and used as described by the manufacturer's instructions.

The medical device in this study is already on the market and is manufactured by Xiros Ltd.

The Pitch-Patch is a single-use polyester prosthesis available in two sizes (30x20mm and 35x25mm). It is reinforced around the perimeter and around each eyelet to provide strength and stability to the device and repair.

The study will collect data on patients who meet the entry criteria and have received the device.

This is a single-armed study, meaning all patients will have a Pitch-Patch. The total length of the is expected to be 3 years.

A minimum of 37 patients will be enrolled into the study. Patients will be enrolled at a study specific follow up visit 2-2.5 years after implant, and data for baseline and other time points prior to 2 years (3month, 6month, and 1 year post surgery) will be collected retrospectively from medical records if available.

DETAILED DESCRIPTION:
This is a clinical investigation study with both a prospective and retrospective study design. It will verify the long-term safety and performance of the Pitch-Patch when implanted to reinforce partially repairable rotator cuff tears and used as described by the manufacturer's instructions.

The medical device in this study is already on the market and is manufactured by Xiros Ltd.

The Pitch-Patch is a single-use polyester prosthesis available in two sizes (30x20mm and 35x25mm). It is reinforced around the perimeter and around each eyelet to provide strength and stability to the device and repair.

The study will collect data on patients who meet the entry criteria and have received the device.

This is a single-armed study, meaning all patients will have a Pitch-Patch. The total length of the is expected to be 3 years.

A minimum of 37 patients will be enrolled into the study. Patients will be enrolled at a study specific follow up visit 2-2.5 years after implant, and data for baseline and other time points prior to 2 years (3month, 6month, and 1 year post surgery) will be collected retrospectively from medical records if available.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been treated using a Pitch-Patch device for augmentation or reinforcement of the rotator cuff 2-2.5years prior to enrolment.
* Patient has a baseline Constant Murley Score (CMS), assessed within 30 days prior to implantation of the device.
* Patient must be 16 years old or above.
* Patient is willing to participate in the study, and having been informed of the nature of the study, has provided written informed consent as approved by the Ethics Committee (EC).

Exclusion Criteria:

- The Pitch-Patch has been used outside its intended use.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rotator cuff tear treated with Pitch-Patch for augmentation or reinforcement of the rotator cuff.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Constant Murley Score (CMS) | 2 years
  The primary performance endpoint is the change in the CMS from baseline (if available) and between post-surgery timepoints up to at least 2 years after surgery.
  CMS comprises of 4 parts: Pain reported by the patient (max 15 points), activities of daily living reported by patient (max 20 points), range of movement assess by the examiner (max 40 points), and strength assessed by the examiner (max 25 points).
  Scores range from 0 to 100. Better functioning shoulders will have a greater number of points, up to a maximum of 100 points.
Device Related or Procedure Related Adverse Events | 2 years
  Device related and/ or procedure related adverse events up to at least 2 years after surgery

SECONDARY OUTCOMES:
Re-tear Rate | 2 years
  Number of re-tear events as assessed by radiographical imaging (e.g., MRI, Ultrasound)
Constant Murley Score (subscale) | 2 years
  Change in CMS subscale scores (pain, activities of daily living, strength, and range of movement) from baseline and between post-surgery timepoints.
  CMS subscales: Pain reported by the patient (max 15 points), activities of daily living reported by patient (max 20 points), range of movement assess by the examiner (max 40 points), and strength assessed by the examiner (max 25 points).
  The higher the score, the higher the shoulder function.
Normal Daily Work/ Normal Recreational Activities | 2 years
  Ability to perform normal daily work and normal recreational activities measured by CMS post-surgery.
  A subscale for Constant Murley Score, reported by the patient. Points range from 0-20, the higher the score, the higher the ability to perform normal daily work/ recreational activities.
Tegner Score | 2 years
  Change in Tegner Score from pre-injury and pre-surgery to post-surgery and between post-surgery timepoints.
  The Tegner activity is a scale to identify graded level of activity of a patient. The scale ranges from 0 (very low level of activity) to 10 (extremely active). A score greater than 6 is only achievable with participation in sport.
Subjective Shoulder Value | 2 years
  Change in Subjective Shoulder Value (SSV) score from baseline and between post-surgery timepoints.
  SSV is measured on a percentage scale from 0% to 100%, with a higher percentage reflecting a subjective feel of a normal shoulder.
Tissue Integration into the Pitch Patch | 2 years
  Tissue integration into the Pitch Patch will be assessed up to the 2 year time point and categorised into 'yes' or 'no' by the examiner. Tissue integration can be assessed from the following:
  * Radiological data
  * Histological data
  * Photographic data

IPD SHARING:
Plan to Share IPD: No